CLINICAL TRIAL: NCT01300533
Title: A Phase 1 Open Label, Safety, Pharmacokinetic and Pharmacodynamic Dose Escalation Study of BIND-014 (Docetaxel Nanoparticles for Injectable Suspension), Given by Intravenous Infusion to Patients With Advanced or Metastatic Cancer
Brief Title: A Study of BIND-014 Given to Patients With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BIND Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIND-014-001
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Cancer; Cancer; Solid Tumors
Keywords: Cancer; Neoplasms; Solid Tumor; Ovarian Cancer; Lung Cancer; Non-Small Cell Lung Cancer; Pancreatic Cancer; Breast Cancer; Endometrial Cancer; Melanoma; Prostate Cancer; Skin Cancer; Head and Neck Cancer; Solid Malignancies
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Breast Neoplasms; Endometrial Neoplasms; Melanoma; Prostatic Neoplasms; Skin Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: BIND-014

SUMMARY:
The goal of this Phase 1 clinical research study is to find the highest safe dose of BIND-014 that can be given in the treatment of patients with advanced or metastatic cancer.

DETAILED DESCRIPTION:
The study is designed to explore the safety, tolerability, pharmacokinetics and pharmacodynamics of BIND-014 and define a recommended Phase 2 dose of BIND-014.

All cycles of therapy will consist of the patient taking BIND-014 intravenously once every three weeks or weekly for three out of four weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form. (ICF)
2. At least 18 years old.
3. Patients with histologically or cytologically confirmed advanced or metastatic cancer for which no standard or curative therapy exists.
4. Measurable or evaluable disease per RECIST version 1.1.
5. Eastern Cooperative Oncology Group Performance Status (ECOG) of 0 or 1.
6. Life expectancy of greater than 12 weeks.
7. Female subjects are eligible to enter and participate in the study if they are of:

   1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any woman who:

      * Has had a hysterectomy, or
      * Has had a bilateral oophorectomy (ovariectomy), or
      * Has had a bilateral tubal ligation, or
      * Is post-menopausal (demonstrated total cessation of menses for at least 1 year).
   2. Childbearing (CB) potential, as long as they have a negative serum pregnancy test at screening and at follow-up, and agrees to one of the following:

      * Use an intrauterine device (IUD) with a documented failure rate of less than 1% per year.
      * Use double barrier contraception method defined as condom with spermicidal jelly, foam, suppository, or film; OR diaphragm with spermicide; OR male condom and diaphragm.
      * The woman's sole male sexual partner is a vasectomized male who is sterile prior to the subject's entry into this study.

Exclusion Criteria:

1. Brain metastases or spinal cord compression, unless treatment was completed at least 4 weeks before entry, and stable without steroid treatment for at least 4 weeks.
2. Inadequate bone marrow reserve as demonstrated by an absolute neutrophil count (ANC) < 1.5 x 10^9/L or platelet count < 100 x 10^9/L (cannot be post-transfusion) or hemoglobin < 9 g/dL (can be post-transfusion).
3. Serum bilirubin > 1.2 times the upper limit of normal (ULN).
4. An alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level > 1.5 x ULN with alkaline phosphatase > 2.5 x ULN.
5. Serum creatinine > 1.5 x ULN or a creatinine clearance of < 50 mL/min calculated by Cockcroft-Gault.
6. Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, cardiac [including life-threatening arrhythmias], hepatic, or renal disease).
7. Unresolved toxicity ≥ Common Toxicity Criteria (CTC) grade 2 from previous anti-cancer therapy except alopecia (if applicable) unless agreed that the patient can be entered after discussion with the Medical Monitor.
8. QTc prolongation defined as a QTc with Framingham correction greater than or equal to 470 ms or a prior history of arrhythmias or significant electrocardiogram (ECG) abnormalities. Certain conditions are acceptable (e.g., controlled atrial fibrillation) if agreed to by Medical Monitor.
9. Participation in a study of an investigational agent within 30 days prior to screening.
10. Having received treatment for their cancer (including chemotherapy, surgery and/or radiation) within the 30 days prior to screening.
11. Pregnant or breast-feeding females.
12. Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study (and for up to 26 weeks after the last dose of investigational product) in such a manner that the risk of pregnancy is minimized
13. Peritoneal or pleural effusions requiring a tap more frequently than every 14 days.
14. Any concurrent condition which, in the Investigator's opinion, makes it undesirable for the subject to participate in this study or which would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To assess the dose limiting toxicities (DLTs) of BIND-014 when on day 1 of a 21-day cycle or when given on day 1, 8 and 15 of a 28-day cycle.
  This information will be used to determine the maximum tolerated dose (MTD) of BIND-014 when given weekly or three weeks.

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of BIND-014 following an IV infusion. | First two cycles of BIND-014
  Pharmacokinetic parameters such as time to peak concentration (Tmax), peak concentration (Cmax), minimum concentration (Cmin), volume of distribution (Vd), half life (t1/2), total body clearance (CL) and area under the concentration-time curve (AUC) will be determined for each patient using plasma concentration data.
To assess any preliminary evidence of anti-tumor activity observed with BIND-014. | 18 months
To assess changes in serum tumor markers when appropriate. | 18 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Investigational Site #01, Scottsdale, Arizona
  - Investigational Site #02, Greenbrae, California
  - Investigational Site #04, Los Angeles, California
  - Investigational Site #06, Fort Meyers, Florida
  - Investigational Site #03, Detriot, Michigan
  - Investigational Site #05, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
http://clincancerres.aacrjournals.org/content/early/2016/02/04/1078-0432.CCR-15-2548.full.pdf+html